CLINICAL TRIAL: NCT00104884
Title: Phase II Trial of Depsipeptide (NSC 630176) in Advanced Malignant Melanoma
Brief Title: FR901228 in Treating Patients With Unresectable Stage III or Stage IV Malignant Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated on May 17, 2006 due to slow accrual.
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000415355; U10CA021115 (NIH); E1603 (Other: ECOG-ACRIN Cancer Research Group)
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Results first posted 2016-03-02 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Malignant Melanoma; Melanoma
Keywords: stage III melanoma; stage IV melanoma; Depsipeptide
MeSH Terms: conditions — Melanoma | interventions — Depsipeptides; romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Depsipeptide (Experimental): Depsipeptide is administered as a 4-hour IV infusion weekly in doses of 13 mg/m^2 for 3 weeks. Repeat cycle every 28 days until unacceptable toxicity or disease progression.
  Interventions: Drug: Depsipeptide

INTERVENTIONS:
Drug: Depsipeptide — Given IV
  Other Names: FR901228; FK228

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as FR901228, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well FR901228 works in treating patients with unresectable stage III or stage IV malignant melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with unresectable stage III or stage IV malignant melanoma treated with FR901228 (depsipeptide).

Secondary

* Determine the progression-free and overall survival of patients treated with this drug.
* Determine the toxicity profile of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive FR901228 (depsipeptide) intravenously (IV) over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 22-40 patients will be accrued for this study within 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Stage III unresectable or American Joint Committee on Cancer (AJCC) stage IV cutaneous, mucosal, ocular, or unknown primary melanoma with measurable disease by physical examination or imaging studies.
* Palpable cutaneous or nodal metastases suitable for punch, trucut, or similar biopsy if the patient agrees.
* Normal electrocardiogram (EKG)
* Left ventricular ejection fraction (LVEF) > 40% by Multi Gated Acquisition Scan (MUGA)
* Corrected QT (QTc) < 500 msec
* Age greater than or equal to 18
* Negative pregnancy test
* Fertile patients must use effective contraception
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2
* Normal organ and marrow function
* Patients on hydrochorthiazide should be switched to a potassium-sparing diuretic or another antihypertensive
* At least 4 weeks since prior radiotherapy
* Patients with cardiac hypertrophy may be enrolled but should be carefully monitored.

Exclusion Criteria:

* Prior FR901228 (depsipeptide)
* Prior chemotherapy
* Other concurrent chemotherapy
* Active central nervous system (CNS) metastases by brain computed tomography (CT) scan or magnetic resonance imaging (MRI)
* History of coronary atherosclerotic heart disease
* History of myocardial infarction
* History of congestive heart failure
* Non-melanoma malignancy within the past 5 years except carcinoma in situ or squamous cell or basal cell skin cancer
* Pregnant or nursing women
* Conditions that in the opinion of the investigator would interfere with the ability of the patient to complete this protocol
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Depsipeptide
* Co-medication with an agent that causes QTc prolongation
* Human immunodeficiency virus (HIV) positive patients receiving combination anti-retroviral therapy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements
* Concurrent radiotherapy
* Left ventricular hypertrophy (LVH) on their baseline EKG tracing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2005-10-04 (Actual); Primary Completion 2006-05 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Lawson, MD, Study Chair — Emory University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on January 11, 2005, accrued its first patient on October 4, 2005, and terminated on May 17, 2006 due to slow accrual. Four patients were enrolled.
Period: Overall Study
Arm/Group | Depsipeptide
Started | 4
Completed | 0
Not Completed | 4
Not completed — Disease progression | 4

BASELINE CHARACTERISTICS:
Population: All enrolled patients
Arm/Group | Depsipeptide
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 53.5 [51 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Response to Depsipeptide
Description: Response is evaluated using Solid Tumor Response Criteria (RECIST) and defined as either complete repose (CR) or partial response (PR).
  Per RECIST criteria, CR = disappearance of all target and nontarget lesions; PR = at least 30% decrease in the sum of the longest diameters of target lesions from baseline, and persistence of one or more non-target lesion(s) and/or the maintenance of tumor marker level above the normal limits.
Time Frame: Assessed every 3 months if patient is < 2 years from study entry; every 6 months if patient is 2 - 3 years from study entry, up to 3 years
Population: The study was terminated early due to slow accrual with final accrual of 4 patients. There are no plans to conduct a formal analysis for any outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Depsipeptide
Number analyzed (Participants) | 4
percentage of participants | NA [NA to NA] — The study was terminated early due to slow accrual with final accrual of 4 patients. There are no plans to conduct a formal analysis for any outcome measure.

ADVERSE EVENTS:
Time Frame: Assessed every 4 weeks while on treatment and for 30 days after the end of treatment
Description: Submission of late adverse events is required at follow-up visits up to 3 years .
Arm/Group | Depsipeptide
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Depsipeptide (N=4)
Hypocalcemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Depsipeptide (N=4)
Anemia (Blood and lymphatic system disorders) | 3
Platelets decreased (Investigations) | 2
Fatigue (General disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Infection w/ unk ANC urinary tract NOS (Infections and infestations) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Alkaline phosphatase increased (Investigations) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 2
Creatinine increased (Investigations) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less